CLINICAL TRIAL: NCT03652038
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, 3-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TD-8236 by Inhalation of Single Ascending Doses in Healthy Subjects (Part A) and Multiple Ascending Doses in Subjects With Stable, Mild Asthma (Part B), and Stable, Moderate-to-Severe Asthma (Part C)
Brief Title: Single and Multiple Ascending Dose Study of TD-8236 by Inhalation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0175; 2018-001260-38 (EudraCT Number)
Record Dates: First submitted 2018-08-20; First posted 2018-08-29 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Asthma
Keywords: Single ascending dose; SAD; Multiple ascending dose; MAD; Phase 1; first-in-human; TD-8236; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- TD-8236 for SAD (Part A) (Experimental): 6 out of 8 subjects per cohort (up to 5 cohorts) will be randomized to receive TD-8236
  Interventions: Drug: TD-8236
- Placebo for SAD (Part A) (Placebo Comparator): 2 out of 8 subjects per cohort (up to 5 cohorts) will be randomized to receive placebo
  Interventions: Drug: Placebo
- TD-8236 for MAD (Part B) (Experimental): 6 out of 8 subjects per cohort (up to 6 cohorts) will be randomized to receive TD-8236.
  Interventions: Drug: TD-8236
- Placebo for MAD (Part B) (Placebo Comparator): 2 out of 8 subjects per cohort (up to 6 cohorts) will be randomized to receive placebo.
  Interventions: Drug: Placebo
- TD-8236 for Biomarker (Part C) (Experimental): 8 subjects in each of 2 biomarker cohorts will be randomized to receive TD-8236.
  Interventions: Drug: TD-8236
- Placebo for Biomarker (Part C) (Placebo Comparator): 8 subjects in 1 biomarker cohort will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-8236 — Study drug to be administered via inhaler device
  Arms: TD-8236 for Biomarker (Part C); TD-8236 for MAD (Part B); TD-8236 for SAD (Part A)
Drug: Placebo — Placebo to be administered via inhaler device
  Arms: Placebo for Biomarker (Part C); Placebo for MAD (Part B); Placebo for SAD (Part A)

SUMMARY:
This is a Phase 1, randomized, double-blinded, placebo controlled study. The study consists of 3 parts: Part A is a single ascending dose (SAD) study in healthy subjects, Part B is a multiple ascending dose (MAD) study in subjects with stable, mild asthma, and Part C (Biomarker) is a multiple dose study in subjects with stable, moderate-to-severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 60 years old
* Willing and able to give informed consent and comply with the study
* Body mass index (BMI) 18 to 32 kg/m2 and weighs at least 50 kg
* Women of child bearing potential must have a negative pregnancy test and use a highly efficient birth control method
* Pre-bronchodilator FEV ≥ 70% predicted for MAD cohorts and >40% predicted for biomarker cohorts
* Treatment with inhaled corticosteroids with or without long acting beta agonists
* Additional inclusion criteria apply

Exclusion Criteria:

* Positive for hepatitis A, B or C, HIV or tuberculosis
* Clinically significant abnormalities of laboratory evaluations
* Have abnormal ECG measurements
* Any sign of respiratory tract infection within 6 weeks of screening
* Have a current bacterial, parasitic, fungal or viral infection
* Uses or have used tobacco or nicotine-containing products within 6 months prior to screening
* Additional exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SAD of TD-8236 by assessing the number, severity and type of treatment emergent adverse events | Day 1 through Day 8
To assess the safety and tolerability of MAD of TD-8236 by assessing the number, severity and type of treatment emergent adverse events | Day 1 through Day 14

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of TD-8236 when given as a Single Ascending Dose (SAD): Area under the plasma concentration-time curve (AUC) | Day 1 through Day 4
  Multiple PK variables of TD-8236 will be assessed during SAD and may include, but are not limited to:
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-8236 when given as a Single Ascending Dose (SAD): Maximum observed concentration (Cmax) | Day 1 through Day 4
  Multiple PK variables of TD-8236 will be assessed during SAD and may include, but are not limited to:
  Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-8236 when given as a Single Ascending Dose (SAD): Time to reach maximum observed concentration (Tmax) | Day 1 through Day 4
  Multiple PK variables of TD-8236 will be assessed during SAD and may include, but are not limited to:
  Time to reach maximum observed concentration (Tmax)
Pharmacokinetics (PK) of TD-8236 when given as a Multiple Ascending Dose (MAD): Area under the plasma concentration-time curve (AUC) | Day 1 through Day 9
  Multiple PK variables of TD-8236 will be assessed during MAD and may include, but are not limited to:
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-8236 when given as a Multiple Ascending Dose (MAD): Maximum observed concentration (Cmax) | Day 1 through Day 9
  Multiple PK variables of TD-8236 will be assessed during MAD and may include, but are not limited to:
  Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-8236 when given as a Multiple Ascending Dose (MAD): Time to reach maximum observed concentration (Tmax) | Day 1 through Day 9
  Multiple PK variables of TD-8236 will be assessed during MAD and may include, but are not limited to:
  Time to reach maximum observed concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (2):
- United Kingdom (2):
  - Theravance Biopharma Investigational Site, Manchester, England
  - Theravance Biopharma Investigational Site, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.